CLINICAL TRIAL: NCT06108115
Title: Smartphone-Based Intervention for Sleep Disturbance in Individuals Recovering From Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthRhythms, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0799011810000
Record Dates: First submitted 2023-09-27; First posted 2023-10-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Abuse With Alcohol-Induced Sleep Disorder; Alcohol Use Disorder (AUD); Sleep Disorder; Sleep Disturbance
MeSH Terms: conditions — Alcoholism; Sleep Wake Disorders; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: CueToSleep (Full Intervention Package) (Experimental): Individuals will be randomly allocated to receive the full Health Rhythms package (CueToSleep) program on their smartphones. The package includes 24/7 behavioral sensing from the participant's smartphone using the global positioning system, accelerometer, and screen on/off state, as well as a series of psychoeducational learning screens about the relationship among alcohol, mood disturbance and sleep, and personalized suggestions for behavior change to improve sleep that will be sent to the participant every 3 to 4 days. These suggestions will be based on behaviors indicated by the individual participant's sensor data over the previous 3 to 4 days.
  Interventions: Behavioral: CueToSleep (Full Intervention Package)
- Measure (Behavioral Sensing Only) (No Intervention): Individuals will only be monitored using the passive sensing capabilities of the Full Intervention Package on their smartphones. These participants will not receive psychoeducational learning screens or behavior change suggestions.

INTERVENTIONS:
Behavioral: CueToSleep (Full Intervention Package) — Individuals will be randomly allocated to receive the full Health Rhythms package (CueToSleep) program on their smartphones. The package includes 24/7 behavioral sensing from the participant's smartphone using the global positioning system, accelerometer, and screen on/off state, as well as a series of psychoeducational learning screens about the relationship among alcohol, mood disturbance and sleep, and personalized suggestions for behavior change to improve sleep that will be sent to the participant every 3 to 4 days. These suggestions will be based on behaviors indicated by the individual participant's sensor data over the previous 3 to 4 days.
  Arms: Behavioral: CueToSleep (Full Intervention Package)

SUMMARY:
In order to assess the efficacy of the rhythm stabilization component of Health Rhythms' product in addressing sleep problems, investigators will recruit 128 outpatients over the age of 18, who are in early recovery (at least 2 weeks but no more than 6 months) from Alcohol Use Disorder (AUDIT-C score >4) and are experiencing sleep problems (ISI score >/= 10). 64 of these individuals will be randomly allocated to receive the full HealthRhythms package (sensing, trending, and stabilization) on their smartphones, while 64 will be asked to consent to sensing only. The duration of the study will be 14 weeks.

The primary outcome measures of the RCT will be the ISI (Insomnia Severity Index). The investigators hypothesize that those receiving the full package will demonstrate lower levels of sleep disturbance.

DETAILED DESCRIPTION:
We will conduct a 14-week randomized controlled trial (RCT) of CueToSleep (behavioral monitoring via smartphone sensors and phone-based Cognitive Behavior Therapy for Insomnia) versus Measure (smartphone-based monitoring only). The sample will be 128 individuals with alcohol use disorder who have been abstinent for at least two weeks and are experiencing sleep difficulties. Using a block randomization scheme, these individuals will be randomly allocated on a 1:1 basis to the experimental condition (CueToSleep) or to the control condition (Measure). The components of the CueToSleep intervention include: 1) education about sleep and its regulation and sleep hygiene; 2) alcohol withdrawal-specific psychoeducation 3) personalized and context-specific suggestions for behavior change to address sleep problems using data obtained from the monitoring portion of CueToSleep; 4) feedback to the user on his/her progress; 5) feedback from the user about the usefulness of the suggestions; 6) adjustment of recommendations based on progress, adherence and feedback from the user.

The primary outcome is change in sleep difficulties as measured by the Insomnia Severity Index (ISI). The study is powered to detect at least medium Cohen's d effect size for this primary outcome. The secondary outcome of interest is proportion relapsing to heavy drinking (≥4 drinks in a day for women; ≥5 drinks in a day for men). Number of drinks consumed on the previous day will be queried daily via smartphone and relapse to heavy drinking will be determined from these participant self-reports.

For our primary outcome, we will fit a 2-level linear mixed effects model with a random intercept and slope to test for group (experimental vs. control) differences in the slope of ISI scores over 14 weeks. This model will regress repeatedly measured ISI score on week, group, the week by group interaction, and covariates (age, sex, living status, employment status). Secondarily, to allow further flexibility in the trajectory of ISI scores over the course of the study, we will fit a mixed effects model with categorical time, and specific contrasts to test changes from baseline to 14 weeks.

For our secondary outcome, we will fit a cox proportional hazards model to regress time to relapse on group and covariates (age, sex, living status, employment status). This model accounts for participants who are censored due to early dropout from the study. Secondarily, we will use simple non-parametric statistics to compare the proportion relapsing to heavy drinking in each group.

All analyses will use an intent-to-treat (ITT) strategy where all participants are included regardless of adherence to the randomized condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Meets criteria for lifetime alcohol use disorder (AUD), as defined by DSM-5
3. Score >/= 4 on AUDIT-C
4. Reports difficulties with sleep and scores >/= 10 on the Insomnia Severity Index
5. Has been in recovery (abstinent) for >/= 2 weeks, but less than 6 months
6. Ability and willingness to provide informed consent
7. Ability to understand and comprehend consent and protocol documents in English.
8. Uses a smartphone compatible with the app.

Exclusion Criteria:

1. Psychotic mental disorder other than bipolar disorder
2. Current diagnosis of OCD, anorexia/ bulimia eating disorder, or antisocial personality disorder
3. Acute suicidal ideation with plan or intent
4. Meet DSM-5 criteria for current moderate to severe substance use disorder (SUD)
5. Unable to comply with study procedures or protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change from Baseline at 3, 6,10 and 14 weeks
  The Insomnia Severity Index are self-reported perceptions of sleep

SECONDARY OUTCOMES:
Relapse to Heavy Drinking | Daily over the course of 14 weeks
  Patient self report

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, PhD, Principal Investigator — Health Rhythms
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No